CLINICAL TRIAL: NCT00922129
Title: A Prospective Randomized Pilot Study Examining the Role and Effectiveness of Conversion to Sirolimus Versus CNI Reduction in Renal Transplant Patients With Prostate Cancer
Brief Title: Effectiveness of Conversion to Sirolimus Versus Calcineurin Inhibitor (CNI) Reduction in Renal Transplant Patients With Prostate Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study did not start up as planned.
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Dr Anil Kapoor, McMaster Institute of Urology, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-002-09
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: Sirolimus; Calcineurin inhibitor; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sirolimus; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conversion to sirolimus (Experimental)
  Interventions: Drug: Sirolimus (Rapamune)
- Calcineurim inhibitor reduction (Active Comparator)
  Interventions: Drug: Cyclosporin (Neoral) or Tacrolimus (Prograf)

INTERVENTIONS:
Drug: Sirolimus (Rapamune) — Started at 5 mg (Target levels 6-10mg/mL), Daily, PO, 24 months
  Other Names: RAPAMUNE
  Arms: Conversion to sirolimus
Drug: Cyclosporin (Neoral) or Tacrolimus (Prograf) — Cyclosporin: 3-4 mg/kg, BID, PO, 24 months
  Tacrolimus: 0-.038-0.045 mg/kg, BID, PO, 24 months
  Other Names: Cyclosporin: NEORAL; Tacrolimus: PROGRAF
  Arms: Calcineurim inhibitor reduction

SUMMARY:
The purpose of this study is to evaluate the role and effectiveness of conversion to sirolimus versus CNI reduction in renal transplant patients with prostate cancer.

DETAILED DESCRIPTION:
This study is designed to support the optimal use of mTOR-inhibitor by providing data for the safe and effectiveness use with sirolimus. This study will take into account effectiveness aspects such as malignancy-free survival cancer by reducing the overall exposure to calcineurin inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Male patients ≤ 50 years in their post renal transplant follow-up;
* Biopsy confirmed prostate cancer;
* Stable renal function with GFR ≥ 40 mL/min.

Exclusion Criteria:

* Patients with metastatic disease;
* Uncontrolled hyperlipidemia;
* Proteinuria > 500 mg/day;
* Biopsy evidence of acute rejection within the past 3 months;
* Existence of any surgical or medical condition, other than the current transplant, which in the opinion of the investigator might significantly alter the absorption, distribution, metabolism or excretion of study medication;
* Patients with mental illness;
* Inability to cooperate or communicate with the investigator or unable to complete self administered questionnaires.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Malignancy-free survival | Months 3, 9, 15, 21

SECONDARY OUTCOMES:
Renal function as measured by serum creatinine and calculated creatinine clearance (using the formula of Cockcroft-Gault) | Weeks 1, 3, 6, Months 3, 6, 9, 12, 15, 18, 21 and 24
Testosterone levels | Months 6, 12, 18 and 24
Quality of life | Months 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, Principal Investigator — McMaster Institute of Urology, McMaster University
Locations (1):
- McMaster Institute of Urology - St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada